CLINICAL TRIAL: NCT03915951
Title: A Phase 2, Open-label Study of Encorafenib + Binimetinib in Patients With BRAFV600-mutant Non-small Cell Lung Cancer
Brief Title: An Open-label Study of Encorafenib + Binimetinib in Patients With BRAFV600-mutant Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-818-202; C4221008 (Other: Alias Study Number); 2024-515929-28-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; cancer; non-small cell lung cancer; non small cell lung cancer; NSCLC; Encorafenib; Binimetinib; Phase 2; Open Label; BRAF mutation; BRAF V600E; Array; Stage IV NSCLC; Metastatic NSCLC; PDL1; PD-LI; Immunotherapy; First line platinum based chemotherapy; BRAF inhibitor; V600
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Period (Experimental): Study treatment with encorafenib and binimetinib will be self-administered orally without regard to food.
  Patients will receive the following per 28-day (± 3 days) cycle:
  * Encorafenib: 450 mg (6 × 75 mg capsule) once daily (QD)
  * Binimetinib: 45 mg (3 × 15 mg tablet) twice daily (BID)
  Interventions: Drug: encorafenib; Drug: binimetinib

INTERVENTIONS:
Drug: encorafenib — self-administered orally
Drug: binimetinib — self-administered orally

SUMMARY:
This is an open-label, multicenter, non-randomized, Phase 2 study to determine the safety, tolerability and efficacy of encorafenib given in combination with binimetinib in patients with BRAFV600E-mutant metastatic non-small cell lung cancer (NSCLC). Patients who are either treatment-naïve, OR who have received 1) first-line treatment with standard platinum-based chemotherapy, OR 2) first-line treatment with an anti-programmed cell death protein 1 (PD-1)/programmed cell death protein ligand 1 (PD-L1) inhibitor given alone or in combination with platinum-based chemotherapy will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of non-small cell lung cancer (NSCLC) that is currently Stage IV.
* Presence of a BRAFV600E mutation in lung cancer tissue as determined by a local laboratory assay or the presence of other BRAFV600 mutations other than V600E (i.e. K or D) will be considered
* Patients who are either treatment-naïve (e.g., no prior systemic therapy for advanced/metastatic disease), OR who have received 1) first-line platinum-based chemotherapy OR 2) first-line treatment with an anti-programmed cell death protein 1 (PD-1)/ programmed cell death protein ligand 1(PD-L1) inhibitor given alone or in combination with platinum-based chemotherapy.
* Presence of measurable disease based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Eastern Cooperation Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow function characterized by the following at screening:

  * absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
  * Platelets ≥ 100 × 10⁹/L;
  * Hemoglobin ≥ 8.5 g/dL (with or without blood transfusions).
* Adequate hepatic and renal function characterized by the following at screening:

  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5 × ULN in presence of liver metastases; Serum creatinine ≤ 1.5 × ULN; or calculated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula; or estimated glomerular filtration rate > 50 mL/min/1.73m².

Key Exclusion Criteria:

* Patients who have documentation of any of the following:

  * epidermal growth factor receptor (EGFR) mutation
  * anaplastic lymphoma kinase (ALK) fusion oncogene or
  * ROS1 rearrangement
* Patients who have received more than 1 prior line of systemic therapy in the advanced/metastatic setting.
* Previous treatment with any BRAF inhibitor (e.g., dabrafenib, vemurafenib, XL281/BMS-908662, etc.), or any mitogen-activated protein kinase (MEK) inhibitor (e.g., trametinib, cobimetinib, selumetinib, RDEA119, etc.) prior to screening and enrollment.
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease.
* Concurrent neuromuscular disorder that is associated with the potential of elevated creatine (phospho)kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Patients with symptomatic brain metastasis, leptomeningeal disease or other active central nervous system (CNS) metastases are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2025-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (135):
- United States (104):
  - Yuma Regional Medical Center Cancer Center, Yuma, Arizona
  - Yuma Regional Medical Center Ophthalmology, Yuma, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - UCLA Stein Eye Center Santa Monica (OPH), Santa Monica, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Florida Cancer Specialist, Altamonte Springs, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialist, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialist, Clearwater, Florida
  - Florida Cancer Specialists, Fleming Island, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialist, Gainesville, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialist, Lecanto, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialist, Ocala, Florida
  - Florida Cancer Specialist, Orange City, Florida
  - Florida Cancer Specialist, Orlando, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialist, St. Petersburg, Florida
  - Florida Cancer Specialists PAN - SCRI - PPDS, Tallahassee, Florida
  - Florida Cancer Specialist, Tampa, Florida
  - Florida Cancer Specialist, Tavares, Florida
  - Florida Cancer Specialist, The Villages, Florida
  - Florida Cancer Specialist, Trinity, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Winship Cancer Institute @ Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Winship Cancer Institute @ Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Winship Cancer Institute @ Emory Johns Creek Hospital, Johns Creek, Georgia
  - MidAmerica Division, Inc. c/o Menorah Medical Center, Overland Park, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Johns Hopkins Wilmer Eye Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston (OCB), Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center/East, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - MidAmerica Division, Inc. c/o Centerpoint Medical Center, Independence, Missouri
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Metropolitan Eye Care, Paramus, New Jersey
  - Memorial Sloan Kettering Cancer Center David H Koch Center for Cancer Care, New York, New York
  - Weill Cornell Eye Associates, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Ohio State CarePoint East, Columbus, Ohio
  - The Ohio State University East Hospital, Columbus, Ohio
  - The Ohio State University Hospital, Columbus, Ohio
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - The Ohio State University Medical Center - Thoracic Oncology Clinic, Columbus, Ohio
  - Ohio State Eye and Ear Institute, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Cancer, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - Ohio State CarePoint Gahanna, Gahanna, Ohio
  - Ohio State Outpatient Care Lewis Center, Lewis Center, Ohio
  - The Ohio State University East Hospital Ohio State Outpatient Care New Albany, Westerville, Ohio
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Cancer Institute Newberg Clinic, Newberg, Oregon
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hillman Cancer Center - Arnold Palmer - Mt View, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center Monroeville, Monroeville, Pennsylvania
  - UPMC Eye Center, Eye and Ear Institute, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant (HOA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant (OHA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - Weaver Eye Associates, York, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - WellSpan Oncology Research, York, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Cleveland, Tennessee
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hendersonville, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Houston Eye Associates - Gramercy Location, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Research & Clinical Development, Houston, Texas
  - Eye associates Northwest, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Italy (9):
  - Unita Operativa Radiologia, Milan, Lombardy
  - Clinica Oculistica II, 2° Policlinico Federico II, Napli, Napli
  - S.S.D. Oncologia Polmonare, Orbassano, Torino
  - SCDU Radiodiagnostica e S.S. Medicina Nucleare, Orbassano, Torino
  - Dermatologia Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Torino, TO
  - UO di Oftalmologia- Azienda Ospedaliero Universitaria Di Bologna, Bologna
  - UOC di Anatomia Patologica- Azienda Ospedaliero Universitaria Di Bo logna, Bologna
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Giovanni Pascale, Napoli
- Netherlands (4):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - OLVG, locatie Oost; Ophthalmology department, Amsterdam
  - Ophthalmology department, Groningen
  - University Medical Center Groningen, Groningen
- Samsung Medical Center - PPDS, Seoul, South Korea
- Spain (17):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Málaga
  - Hospital Clinic de Barcelona, Badalona
  - Hospital del Mar, Barcelona
  - CETIR Centro Medico Teknon, Barcelona
  - Hospital Quiron Salud Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Grupo Cardiologico Corpal (Hospital de la Cruz Roja), Córdoba
  - Hospital Universitario Reina Sofia, Córdoba
  - Cetir, Esplugues de Llobregat
  - lnstitut Catala d'Oncologia_L'Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Hospitalario Integral Privado (CHIP), Málaga
  - CERCO, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Johnson ML, Smit EF, Felip E, Ramalingam SS, Ahn MJ, Tsao A, Johnson BE, Offin M, Hussein M, Dagogo-Jack I, Goldman JW, Clarke JM, Negrao MV, Sanborn RE, Morgensztern D, Usari T, Wilner K, Alejandro L, Rifi N, Zhang X, Riely GJ. Updated Overall Survival Analysis From the Phase II PHAROS Study of Encorafenib Plus Binimetinib in Patients With BRAF V600E-Mutant Metastatic Non-Small Cell Lung Cancer. J Clin Oncol. 2025 Dec 10;43(35):3706-3713. doi: 10.1200/JCO-25-02023. Epub 2025 Oct 19. PMID 41109959
- [Derived] Riely GJ, Ahn MJ, Clarke JM, Dagogo-Jack I, Esper R, Felip E, Gelsomino F, Goldman JW, Hussein M, Johnson M, Marrone KA, Morgensztern D, Nadal E, Negrao MV, Offin M, Provencio M, Ramalingam SS, Roof L, Sanborn RE, Smit EF, Tsao A, Usari T, Alcasid A, Wilner K, Tonkovyd S, Zhang X, Johnson BE. Updated Efficacy and Safety From the Phase 2 PHAROS Study of Encorafenib Plus Binimetinib in Patients With BRAF V600E-Mutant Metastatic NSCLC-A Brief Report. J Thorac Oncol. 2025 Oct;20(10):1538-1547. doi: 10.1016/j.jtho.2025.05.023. Epub 2025 Jun 4. PMID 40480428
- [Derived] Riely GJ, Smit EF, Ahn MJ, Felip E, Ramalingam SS, Tsao A, Johnson M, Gelsomino F, Esper R, Nadal E, Offin M, Provencio M, Clarke J, Hussain M, Otterson GA, Dagogo-Jack I, Goldman JW, Morgensztern D, Alcasid A, Usari T, Wissel P, Wilner K, Pathan N, Tonkovyd S, Johnson BE. Phase II, Open-Label Study of Encorafenib Plus Binimetinib in Patients With BRAFV600-Mutant Metastatic Non-Small-Cell Lung Cancer. J Clin Oncol. 2023 Jul 20;41(21):3700-3711. doi: 10.1200/JCO.23.00774. Epub 2023 Jun 4. PMID 37270692
- [Derived] Riely GJ, Ahn MJ, Felip E, Ramalingam SS, Smit EF, Tsao AS, Alcasid A, Usari T, Wissel PS, Wilner KD, Johnson BE. Encorafenib plus binimetinib in patients with BRAFV600-mutant non-small cell lung cancer: phase II PHAROS study design. Future Oncol. 2022 Mar;18(7):781-791. doi: 10.2217/fon-2021-1250. Epub 2021 Dec 17. PMID 34918546
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-818-202

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment-Naive: Treatment-naïve participants with BRAF V600E-mutant metastatic NSCLC were enrolled to receive encorafenib 450 mg QD and binimetinib 45 mg BID in 28-day (±3 days) cycles and continued until the participants met the protocol-defined criteria for treatment withdrawal.
- Previously Treated: Patients who had received 1) first-line treatment with standard platinum-based chemotherapy, or 2) first-line treatment with an anti-PD-1/PD-L1 inhibitor given alone, or in combination with platinum-based chemotherapy, or in combination with immunotherapy (eg, ipilimumab) with or without platinum-based chemotherapy were enrolled to receive encorafenib 450 mg QD and binimetinib 45 mg BID was to be administered in 28-day (±3 days) cycles and continued until the participants met the protocol-defined criteria for treatment withdrawal.
Period: Overall Study
Arm/Group | Treatment-Naive | Previously Treated
Started | 59 | 39
Completed | 0 | 0
Not Completed | 59 | 39
Not completed — As of the PCD data-cut, 33 participants remained on-treatment. | 25 | 8
Not completed — Adverse Event | 12 | 6
Not completed — Disease progression (radiological) | 17 | 15
Not completed — Disease progression (clinical) | 4 | 1
Not completed — Patient decision | 0 | 4
Not completed — Investigator decision | 0 | 1
Not completed — Consent withdrawn | 1 | 1
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants taking at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Age, Continuous [Median (Full Range); unit: Years] | 68 [47 to 83] | 71 [53 to 86] | 69.5 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 19 | 52
  Male | 26 | 20 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 53 | 33 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Eastern Cooperation Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scoring: Grade 0: Fully active, able to carry on all predisease performance without restriction; Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours; Grade 3: capable of only limited self-care; confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair; Grade 5: dead.
  Participants
    Grade 0 | 19 | 7 | 26
    Grade 1 | 40 | 32 | 72
Smoking Status [Count of Participants; unit: Participants] — Smoking history was collected at Screening by the Investigator or qualified designee.
  Participants
    Current Smoking | 8 | 5 | 13
    Former Smoking | 33 | 23 | 56
    Never Smoking | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response (OR) as Determined by Independent Radiology Review (IRR)
Description: Objective Response Rate (ORR) was defined as the percentage of participants who had achieved a confirmed best overall response (Complete Response [CR] or Partial Response [PR]) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. CR was defined by the disappearance of all non-lymph node target lesions (where all target lesions were recorded with a length of 0 mm, and any pathological lymph nodes [recorded as target lesion] must have reduction in short axis to <10 mm) and complete disappearance of all non-target lesions (where all non-target lesions were marked "Absent", and all lymph nodes must be non-pathological in size [<10 mm in short axis]). PR was defined by a 30% or more decrease in sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. ORR was calculated with the exact 2-sided Clopper-Pearson 95% CI.
Time Frame: From date of the first dose of study intervention until documented progressive disease (PD) or start of new anticancer therapy (up to 36 months)
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive | Previously Treated
Number analyzed (Participants) | 59 | 39
Percentage of Participants | 74.6 [61.6 to 85.0] | 46.2 [30.1 to 62.8]

2. Secondary Outcome: Percentage of Participants With Confirmed Objective Response (OR) by Investigator Assessment
Description: ORR was defined as the percentage of participants who had achieved a confirmed best overall response (CR or PR) per RECIST version 1.1. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. CR was defined by the disappearance of all non-lymph node target lesions (where all target lesions were recorded with a length of 0 mm, and any pathological lymph nodes [recorded as target lesion] must have reduction in short axis to <10 mm) and the complete disappearance of all non-target lesions (where all non-target lesions were marked "Absent", and all lymph nodes must be non-pathological in size [<10 mm in short axis]). PR was defined by a 30% or more decrease in SOD of target lesions, taking as reference the baseline SOD. ORR according to derived investigator assessment was calculated with the exact 2-sided Clopper-Pearson 95% CI.
Time Frame: From date of the first dose of study intervention until documented PD or start of new anticancer therapy (up to 36 months)
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive | Previously Treated
Number analyzed (Participants) | 59 | 39
Percentage of Participants | 62.7 [49.1 to 75.0] | 41.0 [25.6 to 57.9]

3. Secondary Outcome: Duration of Response (DoR) by IRR and Investigator Assessments
Description: DoR, based on IRR and Investigator assessments was defined as the time from the date of the first documented confirmed response (CR or PR) (by IRR and by Investigator, respectively) to the earliest date of disease progression, as determined by Investigator review of radiographic disease assessments and IRR per RECIST version 1.1, or death due to any cause. If a participant with a CR or PR had neither progressed nor died at the time of the analysis cutoff or at the start of any new anticancer therapy, the participant was censored at the date of last adequate tumor assessment. CR was defined by the disappearance of all non-lymph node target lesions and complete disappearance of all non-target lesions. PR was defined by a 30% or more decrease in SOD of target lesions, taking as reference the baseline SOD. DoR was calculated for participants who had achieved a confirmed overall response (CR or PR). The estimate of the DoR survival function was constructed using the Kaplan-Meier method.
Time Frame: From the date of the first confirmed documented response (CR or PR) to the earliest date of disease progression or death due to any cause (up to 36 months)
Reporting Status: Not Posted, anticipated posting 2026-10

4. Secondary Outcome: Disease Control Rate (DCR) by IRR and Investigator Assessments
Description: DCR was defined as the percentage of participants who had achieved a confirmed overall response of CR, PR or stable disease (SD), as determined by Investigator review of radiographic disease assessments and IRR per RECIST version 1.1 after 24 weeks (≥168 days) from the date of first dose of study intervention. CR was defined by the disappearance of all non-lymph node target lesions and complete disappearance of all non-target lesions. PR was defined by a 30% or more decrease in SOD of target lesions, taking as reference the baseline SOD. SD was assigned when neither sufficient shrinkage to qualify for CR or PR, nor sufficient increase to qualify for PD was observed, taking as reference the nadir. DCR was calculated along with the exact 2-sided Clopper-Pearson 95% CI.
Time Frame: After 24 Weeks (≥168 days) from the date of first dose of study intervention
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment-Naive | Previously Treated
Number analyzed (Participants) | 59 | 39
Percentage of Participants
  DCR After 24 Weeks by IRR | 64.4 [50.9 to 76.4] | 41.0 [25.6 to 57.9]
  DCR After 24 Weeks by Investigator Assessment | 67.8 [54.4 to 79.4] | 48.7 [32.4 to 65.2]

5. Secondary Outcome: Progression-free Survival (PFS) by IRR and Investigator Assessments
Description: PFS was defined as the time from the date of first dose of study intervention to the earliest date of disease progression, as determined by IRR and Investigator review of radiographic disease assessments per RECIST version 1.1, or death due to any cause, whichever occurred first. PD was defined by a 20% or more increase in the SOD of target lesions relative to nadir (smallest SOD considering baseline and all assessments prior to the time point under evaluation), with a minimum absolute increase of 5 mm relative to nadir; PD was assigned if any non-target lesion was marked "unequivocal progression". If a participant had not had a PFS event at the time of the analysis cutoff or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment. PFS (months) = [(date of event or censoring - date of first dose) +1]/30.4375. The survival distribution function for PFS was estimated using the Kaplan-Meier method.
Time Frame: From the date of first dose of study drug to the earliest date of disease progression, or death due to any cause (up to 36 months)
Reporting Status: Not Posted, anticipated posting 2026-10

6. Secondary Outcome: Time to Response (TTR) by IRR and Investigator Assessments
Description: TTR based on IRR and Investigator assessments was defined, for participants with an objective response, as the time, in months, from the date of first dose to the first documentation of objective response (CR or PR) which was subsequently confirmed (by IRR and by Investigator, respectively). TTR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: From the date of first dose to the first documentation of confirmed objective response (CR or PR) (up to 36 months)
Population: Analysis population included all participants who received at least 1 dose of study intervention and who had confirmed objective tumor response (CR or PR). Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment-Naive | Previously Treated
Number analyzed (Participants) | 59 | 39
Months
  TTR by IRR: number analyzed (Participants) | 44 | 18
  TTR by IRR | 1.86 [1.1 to 19.1] | 1.74 [1.2 to 7.3]
  TTR by Investigator Assessment: number analyzed (Participants) | 37 | 16
  TTR by Investigator Assessment | 1.84 [1.4 to 14.0] | 1.81 [0.8 to 9.2]

7. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study intervention to the date of death due to any cause. If a death had not been observed by the date of the analysis cutoff, OS was censored at the date of last contact. The survival distribution function for OS was estimated using the Kaplan-Meier method.
Time Frame: The time from the date of first dose of study intervention to the date of death due to any cause (up to 36 months)
Reporting Status: Not Posted, anticipated posting 2026-10

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAE was a treatment-emergent adverse event that occurred during the on-treatment period. The on-treatment period was defined as the time from the first dose date of study intervention to the last dose of study drug administration date (when both drugs were permanently discontinued) +30 days or the earliest date of subsequent anti-cancer drug therapy minus 1 day, whichever occurred first. Relatedness to study intervention was determined by the investigator. The investigator made an assessment of intensity for each AE reported during the study according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03: Grade 3 events = severe AEs; Grade 4 events = life-threatening consequences, urgent intervention indicated; Grade 5 events = death related to AEs.
Time Frame: From the time the participant provided informed consent, through and including a minimum of 30 calendar days, after the last administration of the study intervention, and the safety follow-up visit (30 days [±7 days] after the EOT visit) (up to 36 months)
Population: Safety Analysis Set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Sum of all participants in the Study C4221008 (ARRAY-818-202)
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Participants
  Participants With TEAEs | 59 | 38 | 97
  Participants With Treatment-related TEAEs | 58 | 34 | 92
  Participants with Maximum Grade 3 or 4 TEAEs | 37 | 18 | 55
  Participants with Maximum Treatment-related Grade 3 or 4 TEAEs | 27 | 13 | 40
  Participants With Grade 5 TEAEs | 5 | 7 | 12
  Participants With Treatment-related Grade 5 TEAEs | 1 | 0 | 1

9. Secondary Outcome: Number of Participants With Shifts From Grade ≤2 at Baseline to Grade 3 or 4 at Post-baseline in Hematology Laboratory Test Values Based on CTCAE Grade
Description: Blood and urine samples for the laboratory tests. A central laboratory will perform all clinical laboratory assessments. Baseline was the last available assessment performed prior to the study intervention start date/time.
  Grade 4 was not applicable for the parameters of anemia, hemoglobin increased, leukocytosis and lymphocyte count increased as Grade 4 was not defined for these 4 parameters per CTCAE version 4.03.
Time Frame: Screening, Cycle 1 Day 1, Cycle 2 Day 1 ±3 Days, Day 1 ±3 Days in Subsequent Cycles, End of Treatment (EOT) ±3 Days and Safety Follow-up Visit (30 Days [±7 Days] After the EOT Visit) (Up to 36 Months)
Population: Safety Analysis Set included all participants who received at least 1 dose of study intervention. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Participants
  Anemia - Grade 3: number analyzed (Participants) | 55 | 38 | 93
  Anemia - Grade 3 | 9 | 1 | 10
  Hemoglobin increased - Grade 3: number analyzed (Participants) | 55 | 38 | 93
  Hemoglobin increased - Grade 3 | 0 | 0 | 0
  Leukocytosis - Grade 3: number analyzed (Participants) | 55 | 38 | 93
  Leukocytosis - Grade 3 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 3: number analyzed (Participants) | 54 | 37 | 91
  Lymphocyte count decreased - Grade 3 | 2 | 3 | 5
  Lymphocyte count decreased - Grade 4: number analyzed (Participants) | 54 | 37 | 91
  Lymphocyte count decreased - Grade 4 | 0 | 0 | 0
  Lymphocyte count increased - Grade 3: number analyzed (Participants) | 54 | 37 | 91
  Lymphocyte count increased - Grade 3 | 0 | 0 | 0
  Neutrophil count decreased - Grade 3: number analyzed (Participants) | 54 | 37 | 91
  Neutrophil count decreased - Grade 3 | 1 | 0 | 1
  Neutrophil count decreased - Grade 4: number analyzed (Participants) | 54 | 37 | 91
  Neutrophil count decreased - Grade 4 | 0 | 0 | 0
  Platelet count decreased - Grade 3: number analyzed (Participants) | 55 | 38 | 93
  Platelet count decreased - Grade 3 | 0 | 1 | 1
  Platelet count decreased - Grade 4: number analyzed (Participants) | 55 | 38 | 93
  Platelet count decreased - Grade 4 | 0 | 0 | 0
  White blood cell decreased - Grade 3: number analyzed (Participants) | 55 | 38 | 93
  White blood cell decreased - Grade 3 | 0 | 0 | 0
  White blood cell decreased - Grade 4: number analyzed (Participants) | 55 | 38 | 93
  White blood cell decreased - Grade 4 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Shifts From Grade ≤2 at Baseline to Grade 3 or 4 at Post-baseline in Chemistry Laboratory Test Values Based on CTCAE Grade
Description: Blood and urine samples for the laboratory tests. A central laboratory will perform all clinical laboratory assessments. Baseline was the last available assessment performed prior to the study intervention start date/time.
  Grade 4 was not applicable for the parameters of hyperglycemia and hypoalbuminemia as Grade 4 was not defined for these 2 parameters per CTCAE version 4.03.
Time Frame: Screening, Cycle 1 Day 1, Cycle 2 Day 1 ±3 Days, Day 1 ±3 Days in Subsequent Cycles, EOT ±3 Days and Safety Follow-up Visit (30 Days [±7 Days] After the EOT Visit) (Up to 36 Months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Participants
  Alanine aminotransferase increased - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Alanine aminotransferase increased - Grade 3 | 6 | 2 | 8
  Alanine aminotransferase increased - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Alanine aminotransferase increased - Grade 4 | 0 | 0 | 0
  Alkaline phosphatase increased - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Alkaline phosphatase increased - Grade 3 | 2 | 1 | 3
  Alkaline phosphatase increased - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Alkaline phosphatase increased - Grade 4 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Aspartate aminotransferase increased - Grade 3 | 7 | 2 | 9
  Aspartate aminotransferase increased - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Aspartate aminotransferase increased - Grade 4 | 0 | 0 | 0
  Blood bilirubin increased - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Blood bilirubin increased - Grade 3 | 0 | 0 | 0
  Blood bilirubin increased - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Blood bilirubin increased - Grade 4 | 0 | 0 | 0
  Creatine kinase increased - Grade 3: number analyzed (Participants) | 55 | 36 | 91
  Creatine kinase increased - Grade 3 | 2 | 1 | 3
  Creatine kinase increased - Grade 4: number analyzed (Participants) | 55 | 36 | 91
  Creatine kinase increased - Grade 4 | 0 | 0 | 0
  Creatinine increased - Grade 3: number analyzed (Participants) | 57 | 38 | 95
  Creatinine increased - Grade 3 | 3 | 0 | 3
  Creatinine increased - Grade 4: number analyzed (Participants) | 57 | 38 | 95
  Creatinine increased - Grade 4 | 0 | 0 | 0
  Hypercalcemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypercalcemia - Grade 3 | 1 | 1 | 2
  Hypercalcemia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hypercalcemia - Grade 4 | 0 | 0 | 0
  Hyperglycemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hyperglycemia - Grade 3 | 5 | 1 | 6
  Hyperkalemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hyperkalemia - Grade 3 | 2 | 0 | 2
  Hyperkalemia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hyperkalemia - Grade 4 | 0 | 0 | 0
  Hypermagnesemia - Grade 3: number analyzed (Participants) | 55 | 36 | 91
  Hypermagnesemia - Grade 3 | 0 | 1 | 1
  Hypermagnesemia - Grade 4: number analyzed (Participants) | 55 | 36 | 91
  Hypermagnesemia - Grade 4 | 0 | 0 | 0
  Hypernatremia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypernatremia - Grade 3 | 0 | 0 | 0
  Hypernatremia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hypernatremia - Grade 4 | 0 | 0 | 0
  Hypoalbuminemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypoalbuminemia - Grade 3 | 0 | 0 | 0
  Hypocalcemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypocalcemia - Grade 3 | 0 | 0 | 0
  Hypocalcemia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hypocalcemia - Grade 4 | 2 | 0 | 2
  Hypoglycemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypoglycemia - Grade 3 | 0 | 0 | 0
  Hypoglycemia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hypoglycemia - Grade 4 | 0 | 0 | 0
  Hypokalemia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hypokalemia - Grade 3 | 0 | 1 | 1
  Hypokalemia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hypokalemia - Grade 4 | 0 | 0 | 0
  Hypomagnesemia - Grade 3: number analyzed (Participants) | 55 | 36 | 91
  Hypomagnesemia - Grade 3 | 0 | 0 | 0
  Hypomagnesemia - Grade 4: number analyzed (Participants) | 55 | 36 | 91
  Hypomagnesemia - Grade 4 | 0 | 0 | 0
  Hyponatremia - Grade 3: number analyzed (Participants) | 56 | 38 | 94
  Hyponatremia - Grade 3 | 7 | 2 | 9
  Hyponatremia - Grade 4: number analyzed (Participants) | 56 | 38 | 94
  Hyponatremia - Grade 4 | 0 | 0 | 0
  Hypophosphatemia - Grade 3: number analyzed (Participants) | 55 | 36 | 91
  Hypophosphatemia - Grade 3 | 1 | 0 | 1
  Hypophosphatemia - Grade 4: number analyzed (Participants) | 55 | 36 | 91
  Hypophosphatemia - Grade 4 | 0 | 0 | 0
  Lipase increased - Grade 3: number analyzed (Participants) | 56 | 36 | 92
  Lipase increased - Grade 3 | 8 | 3 | 11
  Lipase increased - Grade 4: number analyzed (Participants) | 56 | 36 | 92
  Lipase increased - Grade 4 | 2 | 0 | 2
  Serum amylase increased - Grade 3: number analyzed (Participants) | 56 | 36 | 92
  Serum amylase increased - Grade 3 | 1 | 0 | 1
  Serum amylase increased - Grade 4: number analyzed (Participants) | 56 | 36 | 92
  Serum amylase increased - Grade 4 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Notable Abnormal Vital Signs
Description: Vital sign measurements were taken before blood collection for laboratory tests or at least 30 minutes after blood collection for laboratory tests, and were measured per institutional standards. Vital sign assessments included temperature, pulse rate, respiratory rate, and blood pressure (assessed in a recumbent, semi recumbent, or sitting position).
  The criteria of notably abnormal vital signs are listed below:
  Systolic blood pressure (mmHg): high: ≥160 mmHg with increase from baseline of ≥20 mmHg; low: ≤90 mmHg with decrease from baseline of ≥20 mmHg.
  Diastolic blood pressure (mmHg): high: ≥100 mmHg with increase from baseline of ≥15 mmHg; low: ≤50 mmHg with decrease from baseline of ≥15 mmHg.
  Pulse rate (bpm): high: ≥120 bpm with increase from baseline of ≥15 bpm; low: ≤50 bpm with decrease from baseline of ≥15 bpm.
  Weight (kg): high: ≥10% increase from baseline; low: ≥20% decrease from baseline.
  Temperature (°C): high: ≥37.5 °C; low: ≤36 °C.
Time Frame: Screening, Cycle 1 Day 1, Cycle 2 Day 1 ±3 Days, Day 1 ±3 Days of Subsequent Cycles, EOT ±3 Days, and Safety Follow-up Visit (30 Days [±7 Days] After the EOT Visit) (Up to 36 Months)
Population: Analysis population included all participants who received at least 1 dose of study intervention and had baseline and post-baseline vital sign values. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Participants
  Systolic blood pressure - high: number analyzed (Participants) | 58 | 38 | 96
  Systolic blood pressure - high | 10 | 4 | 14
  Systolic blood pressure - low: number analyzed (Participants) | 58 | 38 | 96
  Systolic blood pressure - low | 5 | 2 | 7
  Diastolic blood pressure - high: number analyzed (Participants) | 58 | 38 | 96
  Diastolic blood pressure - high | 5 | 1 | 6
  Diastolic blood pressure - low: number analyzed (Participants) | 58 | 38 | 96
  Diastolic blood pressure - low | 2 | 2 | 4
  Pulse rate - high: number analyzed (Participants) | 58 | 38 | 96
  Pulse rate - high | 2 | 6 | 8
  Pulse rate - low: number analyzed (Participants) | 58 | 38 | 96
  Pulse rate - low | 1 | 1 | 2
  Weight - high: number analyzed (Participants) | 57 | 38 | 95
  Weight - high | 17 | 4 | 21
  Weight - low: number analyzed (Participants) | 57 | 38 | 95
  Weight - low | 1 | 0 | 1
  Temperature - high: number analyzed (Participants) | 58 | 38 | 96
  Temperature - high | 8 | 3 | 11
  Temperature - low: number analyzed (Participants) | 58 | 38 | 96
  Temperature - low | 25 | 10 | 35

12. Secondary Outcome: Number of Participants With Notable ECG (QTcF) Values
Description: The QTcF increase from baseline >30/60 msec and new QTcF >450/480/500 msec were defined as clinically notable ECG criteria. Triplicate ECG measurements were obtained. For new abnormal post-baseline values, the table below presents the number of participants with both non-missing baseline and post-baseline values, and baseline values not meeting the criteria. For abnormal changes from baseline, the table below presents the number of participants with both non-missing baseline and post-baseline evaluations. Baseline was defined as the average of the machine-read triplicate ECG measurements taken pre-dose on Day 1. Change from baseline was post-baseline - baseline values.
Time Frame: Screening, Cycle 1 Day 1, Cycle 2 Day 1 ±3 Days, Every 12 Weeks ±7 Days, and EOT ±3 Days (Up to 36 Months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 59 | 39 | 98
Participants
  New QTcF >450 msec: number analyzed (Participants) | 54 | 31 | 85
  New QTcF >450 msec | 12 | 7 | 19
  New QTcF >480 msec: number analyzed (Participants) | 57 | 37 | 94
  New QTcF >480 msec | 5 | 5 | 10
  New QTcF >500 msec: number analyzed (Participants) | 58 | 37 | 95
  New QTcF >500 msec | 1 | 1 | 2
  QTcF Increase from baseline >30 msec: number analyzed (Participants) | 58 | 38 | 96
  QTcF Increase from baseline >30 msec | 20 | 9 | 29
  QTcF Increase from baseline >60 msec: number analyzed (Participants) | 58 | 38 | 96
  QTcF Increase from baseline >60 msec | 3 | 4 | 7

13. Secondary Outcome: Number of Participants With the Worst Post-baseline Left Ventricular Ejection Fraction (LVEF) Values Based on CTCAE Grade
Description: Cardiac ejection fraction was assessed by transthoracic echocardiogram (ECHO) or multigated acquisition (MUGA). Participants who developed signs/symptoms of congestive heart failure (CHF) at any point during the study were required to have an evaluation of LVEF measurements by ECHO or MUGA and were monitored per institutional guidelines.
  Participants were considered as having a LVEF abnormality if the worst post-value was CTCAE Grade 2, 3 or 4 according to the following classification:
  Grade 0: Non-missing value below Grade 2. Grade 2: LVEF between 40% and 50%, inclusive, or absolute change from baseline between -10% and < -20%.
  Grade 3: LVEF between 20% and 39%, inclusive, or absolute change from baseline ≤ -20%.
  Grade 4: LVEF lower than 20%. Baseline was defined as the last available and valid assessment before or on the start date of study intervention.
Time Frame: Screening, Cycle 2 Day 1 ±3 Days, Every 12 Weeks ±7 Days, and EOT ±3 Days (Up to 36 Months)
Population: Analysis Population included all participants who received at least 1 dose of study intervention and had both baseline and post-baseline LVEF values. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naive | Previously Treated | Total
Number analyzed (Participants) | 56 | 33 | 89
Participants
  Grade 0 | 45 | 24 | 69
  Grade 2 | 11 | 7 | 18
  Grade 3 | 0 | 2 | 2
  Grade 4 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the participant provided informed consent, through and including a minimum of 30 calendar days, after the last administration of the study intervention, and the safety follow-up visit (30 days [±7 days] after the EOT visit) (up to 36 months)
Description: Same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both serious and non-serious event during the study. Safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | Treatment-Naive | Previously Treated | Total
All-Cause Mortality (participants affected / at risk) | 5/59 | 7/39 | 12/98
Serious Adverse Events (participants affected / at risk) | 25/59 | 17/39 | 42/98
Other Adverse Events (participants affected / at risk) | 59/59 | 38/39 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=59) | Previously Treated (N=39) | Total (N=98)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 4 | 0 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Disease progression (General disorders) | 2 | 4 | 6
Oedema peripheral (General disorders) | 2 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 2
COVID-19 (Infections and infestations) | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1
Empyema (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=59) | Previously Treated (N=39) | Total (N=98)
Anaemia (Blood and lymphatic system disorders) | 20 | 10 | 30
Vision blurred (Eye disorders) | 14 | 6 | 20
Nausea (Gastrointestinal disorders) | 37 | 19 | 56
Diarrhoea (Gastrointestinal disorders) | 29 | 20 | 49
Vomiting (Gastrointestinal disorders) | 23 | 13 | 36
Constipation (Gastrointestinal disorders) | 18 | 8 | 26
Abdominal pain (Gastrointestinal disorders) | 14 | 6 | 20
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 8
Fatigue (General disorders) | 29 | 16 | 45
Pyrexia (General disorders) | 16 | 6 | 22
Oedema peripheral (General disorders) | 12 | 8 | 20
Asthenia (General disorders) | 7 | 9 | 16
Non-cardiac chest pain (General disorders) | 6 | 2 | 8
Chills (General disorders) | 3 | 3 | 6
Malaise (General disorders) | 5 | 1 | 6
COVID-19 (Infections and infestations) | 5 | 2 | 7
Aspartate aminotransferase increased (Investigations) | 11 | 4 | 15
Blood creatine phosphokinase increased (Investigations) | 10 | 5 | 15
Blood creatinine increased (Investigations) | 8 | 7 | 15
Lipase increased (Investigations) | 11 | 4 | 15
Alanine aminotransferase increased (Investigations) | 10 | 3 | 13
Blood alkaline phosphatase increased (Investigations) | 9 | 2 | 11
Weight increased (Investigations) | 10 | 1 | 11
Ejection fraction decreased (Investigations) | 4 | 4 | 8
SARS-CoV-2 test positive (Investigations) | 4 | 4 | 8
Weight decreased (Investigations) | 6 | 1 | 7
Amylase increased (Investigations) | 4 | 2 | 6
Platelet count decreased (Investigations) | 2 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 12 | 2 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 5 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 1 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 7 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 2 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 7
Dizziness (Nervous system disorders) | 10 | 6 | 16
Headache (Nervous system disorders) | 6 | 4 | 10
Dysgeusia (Nervous system disorders) | 5 | 3 | 8
Paraesthesia (Nervous system disorders) | 5 | 0 | 5
Insomnia (Psychiatric disorders) | 7 | 3 | 10
Pollakiuria (Renal and urinary disorders) | 6 | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 8 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 2 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 3 | 12
Rash (Skin and subcutaneous tissue disorders) | 6 | 5 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3 | 8
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 5 | 1 | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Hypertension (Vascular disorders) | 8 | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03915951/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03915951/SAP_001.pdf